CLINICAL TRIAL: NCT03047642
Title: Validation of Promising Biomarker Assays to Assess Their Diagnostic Performance Characteristics in Africa and Latin America
Brief Title: Validation of Promising Biomarker Assays to Assess Their Diagnostic Performance Characteristics
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Malawi Epidemiology and Intervention Research Unit (Other); Instituto Nacional de Infectologia Evandro Chagas (Unknown); Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Sponsor
Other Study IDs: AFI_01
Record Dates: First submitted 2016-10-10; First posted 2017-02-09 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Febrile Illnesses
Keywords: biomarker; low and middle income countries; fever; antimicrobial resistance; diagnostic
MeSH Terms: conditions — Fever; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of whole blood, plasma, serum and urine are stored to establish a biobank of characterized samples for further development and testing of diagnostic tools for differential diagnosis of multiple febrile diseases in endemic areas.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Malawi febrile patients: Children and adults with fever presenting at the outpatient department
  Interventions: Diagnostic Test: Biomarker assay
- Brazil febrile patients: Children and adults with fever presenting at the outpatient department
  Interventions: Diagnostic Test: Biomarker assay
- Gabon febrile patients: Children with fever or with a recent history of fever presenting at the outpatient department
  Interventions: Diagnostic Test: Biomarker assay

INTERVENTIONS:
Diagnostic Test: Biomarker assay — There is no intervention on the patients but biomarker assays are being evaluated for their performance to distinguish bacterial infection from non-bacterial infections in febrile patients

SUMMARY:
This project aims to evaluate the performance characteristics of rapid tests to differentiate bacterial from non-bacterial infection in febrile adults and children presenting at OPDs (outpatient departments) i.e.("fever triage assays") in three LMICs. The evaluation will include a different commercial biomarker combinations as well as individual biomarkers to assess their individual or combined value in the target population. Markers will be evaluated onsite in ELISA or RDT format, as appropriate. Further, this study aims to contribute to a centralized biobank of well-characterized specimens for use by IVD companies and academic institutions for the development and evaluation of emerging assays.

ELIGIBILITY:
Inclusion Criteria:

Any non-severely ill subject presenting with acute fever defined as: temperature of more than 38°C at initial evaluation of less than 7 days of symptoms at presentation.

Inclusion criteria:

* Children 2-17 years of age
* Adults 18-65 years of age
* Signed written informed consent for study participation. For recruitment purposes, subjects will be classified into two groups, children and adults. For children, age >2 years is the minimum cut-off, based on the amount of blood volume to be obtained in the study. WHO guidelines for allowable blood volume in 24 hours recommend that no more than 1-5% of total blood volume (75-80 ml/kg for older children) be obtained. Applying the average weight of a 2 year old toddler =12 kg, the allowable blood volume to be drawn in 24 hours at 1-5% of the total blood volume is 9.6 - 48 mL .

For minors, caregivers will provide informed consent. Documented assent for children of 12 to 16 years of age will be required for their participation.

Exclusion Criteria:

* Subjects who are felt to be in critical condition (based on clinician assessment or the presence of any general signs of critical illness as defined by WHO guidelines (for children: extensive vomiting, active seizure or recent history of seizures, altered mentation, inability to feed, or any of the severe IMNCI classifications; for adults: impending airway obstruction, central cyanosis, severe respiratory distress, feeble pulse, active seizure or recent history of seizures, or unconsciousness) because the target population for the study is non-severe febrile subjects.
* Subjects can only be enrolled once into the study.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any non-severely ill subject presenting with acute fever defined as: temperature of more than 38°C at initial evaluation of less than 7 days of symptoms at presentation.
  For recruitment purposes, subjects will be classified into two groups:
  * Children 2-17 years of age
  * Adults 18-65 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity to determine bacterial infections compared to clinical and microbiological results aggregated in a study database. | 1year
  Microbiological testing (blood culture positive/negative, malaria pos/neg, S. Tyhpi RDT pos/neg) and clinical assessments of symptoms (respiratory, gastro, no foci) will be recorded and reviewed by a clinical panel upon completion of the study to assign a final category (bacterial or non-bacterial). These categories are used in the evaluation of the biomarker assays to evaluate their performance in differentiating bacterial from non-bacterial infections. Where applicable, the same categories will be used to determine the area under the curve by employing receiver operator characteristics (ROC) analysis of quantitative markers.

CONTACTS AND LOCATIONS:
Locations (3):
- Instituto Nacional de Infectologia Evandro Chagas - Fiocruz (INIEC), Rio de Janeiro, Brazil
- CERMEL, Lambaréné, Gabon
- Karonga Prevention Study, Chilumba, Karonga District, Malawi

IPD SHARING:
Plan to Share IPD: Yes
As appropriate data will be made available to the scientific community and/or commercial partners to support product development activities.

REFERENCES:
- [Derived] Fernandez-Carballo BL, Atzeni M, Escadafal C, Vettoretti M, Geis S, Agnandji ST, Siqueira AM, Malava JK, Banda L, Kabwende AL, Alabi A, Ondo JCB, Massinga-Loembe M, Essone PN, Moreira J, da Rocha Matos A, Caetano BC, Siqueira MM, Bispo de Filippis AM, Dos Santos Ribeiro da Silva EA, Lourenco MCS, Haring J, Gunther A, Jakobi M, Schneiderhan-Marra N, Hoogland C, Brasil P, Pokharel S, Ongarello S, Harris V, Mace A, Lee SJ, Di Camillo B, Dittrich S. Cross-sectional evaluation of host biomarkers for guiding antibiotic use in bacterial and non-bacterial acute febrile illness in low- and middle-income tropical settings. BMJ Open. 2025 Feb 13;15(2):e086912. doi: 10.1136/bmjopen-2024-086912. PMID 39947818